CLINICAL TRIAL: NCT02317679
Title: Treatment of Port-wine Stains by Bosentan in Addition to Pulsed Dye Laser (PDL) in Children or Young Adults Who Previously Failed to Respond to PDL Alone: a Monocentric Pilot Study
Brief Title: Treatment of Resistant Port-wine Stains With Bosentan and Pulsed Dye Laser: a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-PP-10
Record Dates: First submitted 2014-03-21; First posted 2014-12-16 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Port-wine Stains
MeSH Terms: conditions — Port-Wine Stain | interventions — Bosentan; Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosentan and laser (Experimental): Patients with PWS resistant to PDL treatment will be included. A test area of the PWS will be treated by pulsed dye laser (PDL) (λ= 595 nm, 7 mm spot diameter, τp= 1.5 ms, same energy density used at the last session for each subject). The treatment by Bosentan (twice daily :2 mg/kg and maximum 62,5 mg) will be given 1 day before the PDL irradiation (maximum area treated 100 cm2) and continued for 14 days. The clinical improvement of the lesions will be evaluated by comparing standardized pictures, 14 days after the end of the treatment by Bosentan which corresponds to 1 month after the laser PDL irradiation. The evaluation will be realized by 2 independent physicians blinded to the area treated or not. Hemoglobin and SGOT/SGPT will be controlled before and after the treatment by Bosentan.
  Interventions: Drug: Bosentan; Device: Pulsed dye laser (PDL)

INTERVENTIONS:
Drug: Bosentan — Patients with PWS resistant to PDL treatment will be included. The treatment by Bosentan (twice daily :2 mg/kg and maximum 62,5 mg) will be given 1 day before the PDL irradiation (maximum area treated 100 cm2) and continued for 14 days. The clinical improvement of the lesions will be evaluated by comparing standardized pictures, 14 days after the end of the treatment by Bosentan which corresponds to 1 month after the laser PDL irradiation. The evaluation will be realized by 2 independent physicians blinded to the area treated or not. Hemoglobin and SGOT/SGPT will be controlled before and after the treatment by Bosentan.
  Other Names: tracleer
Device: Pulsed dye laser (PDL) — A test area of the PWS will be treated by pulsed dye laser (PDL) (λ= 595 nm, 7 mm spot diameter, τp= 1.5 ms, same energy density used at the last session for each subject).

SUMMARY:
Pulsed dye laser (PDL) is the gold standard treatment for port-wine stains (PWS). However, the outcomes are highly variable due to the new angiogenesis occurring after laser irradiation. Studies suggest that endothelin is involved in the neoangiogenesis that occurred after treatment of port-wine stains by PDL. The main objective of this pilot clinical trial is to evaluate the effectiveness and safety of an inhibitor of endothelin orally taken, the Bosentan, following PDL treatment. Four patients with facial port-wine stain resistant to the PDL treatment will be included. The treatment by Bosentan (2 mg/kg twice daily, maximum 62,5 mg twice daily) will be given one day before the PDL irradiation and continued for 14 days. Only one test area of PWS will be treated with PDL. The primary outcome measure will be an important or complete improvement (Investigator Global Assessment 3 or 4) between treated area and non treated one, 14 days after the end of the treatment which corresponds to one month after the laser PDL session. The evaluation will been performed on standardized pictures by 2 independent physicians blinded to the region treated or not.

DETAILED DESCRIPTION:
Pulsed dye laser (PDL) is the gold standard treatment for port-wine stains (PWS). However, the outcomes are highly variable due to the new angiogenesis occurring after laser irradiation. Studies suggest that endothelin is involved in the neoangiogenesis that occurred after treatment of port-wine stains by PDL . The main objective of this pilot clinical trial is to evaluate the effectiveness and safety of an inhibitor of endothelin orally taken, the Bosentan, following PDL treatment. Four patients with facial port-wine stain resistant to the PDL treatment will be included. The treatment by Bosentan (2 mg/kg twice daily, maximum 62,5 mg twice daily) will be given one day before the PDL irradiation (maximum surface 100 cm²) and continued for 14 days. Only one test area of PWS will be treated with PDL. The primary outcome measure will be an important or complete improvement (Investigator Global Assessment 3 or 4) between treated area and non treated one, 14 days after the end of the treatment which corresponds to one month after the laser PDL session. The evaluation will been performed on standardized pictures by 2 independent physicians blinded to the region treated or not.

ELIGIBILITY:
Inclusion Criteria:

* Children of 7 years old and over or adults aged under 60
* with a resistant port-wine stain after treatment by PDL will be included in this pilot study.
* The agreement of the parents and the child or the patient alone if major will be required.
* Subjects have to be registered to the social security.
* An informed consent will have to be signed by the parents or the patient if of a suitable age or the patient alone if major.
* An efficient contraception will be mandatory if the patient is female and an age to give birth.

Exclusion criteria:

* Hypersensitivity to the Bosentan or to one of its excipients.
* Mild to severe liver disease corresponding to the Child-Pugh Score B or C.
* Serum levels of ASAT and/or ALAT greater three times the upper limit of normal. - Concurrent use of cyclosporine.
* Pregnancy.

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | at 1 month after the start of treatment with bosentan and Pulsed Dye Laser
  The primary outcome measure will be an important or complete improvement (Investigator Global Assessment) between treated area and non treated one, at 1 month after the start of treatment by bosentan and Pulsed Dye Laser

SECONDARY OUTCOMES:
Patient satisfaction | 1 time at 1 month after the start of treatment with bosentan and Pulsed Dye Laser
  The secondary outcome measure will be the satisfaction of the patients (or their parents), or the patient alone if major, about the efficiency and the safety of the treatments at 1 month after the start of treatment by bosentan and Pulsed Dye Laser. A visual analogical scale will be used.
Side effects | 3 times : First time the day of start of bosentan. Second time, one day after the start of treatment with bosentan. The third time, 30 days after the start of treatment with bosentan and pulsed dye laser
  Frequency, severity and occurrence of side effects will be noted.
Satisfaction of the patients of the treatment using visual analogical scale | 1 time at 1 month after the start of treatment by bosentan and Pulsed Dye Laser
  The secondary outcome measure will be the satisfaction of the patients (or their parents), or the patient alone if major, about the safety of the treatments at 1 month after the start of treatment with bosentan and Pulsed Dye Laser

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Thierry, Phd, Principal Investigator — CHU De Nice, Dermatologie, Hôpital de l'archet 151 route de st-antoine de ginestière 06200 nice
Locations (1):
- CHU de Nice - Dermatologie - Hôpital Archet, Nice, Alpes-maritimes, France